CLINICAL TRIAL: NCT04764825
Title: Intraoperative Methadone for Postoperative Pain Management in Spinal Fusion Surgery: a Prospective, Double-blind, Randomised Controlled Trial
Brief Title: Methadone for Spinal Fusion Surgery.
Acronym: METASPINE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to extremely slow inclusion rates.
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 89456049; 2020-004826-47 (EudraCT Number)
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2023-04

CONDITIONS: Pain, Postoperative; Back Pain; Opioid Use; Methadone; Degenerative Spondylolisthesis; Stenosis, Spinal
Keywords: methadone; postoperative; pain; spinalfusion
MeSH Terms: conditions — Pain, Postoperative; Back Pain; Spinal Stenosis; Pain | interventions — Methadone; Morphine

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomisation and study medication will be handled by the hospital pharmacy. All research team members, caregiving clinicians and enrolled patients will be blinded to the study allocation arms and the randomisation list will be concealed until all statistical analyses are made.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Methadone, induction (Experimental): Patients receive methadone 0.15-0.2 mg/kg ideal bodyweight 10 minutes prior to surgery start (Syringe A).
  45 minutes before expected extubation patients will receive saline (syringe B).
  Interventions: Drug: Methadone
- Methadone, end of surgery (Experimental): Patients receive saline 10 minutes prior to surgery start (Syringe A). 45 minutes before expected extubation patients will receive methadone 0.15-0.2 mg/kg ideal bodyweight (syringe B).
  Interventions: Drug: Methadone
- Morphine (Active Comparator): Patients receive saline 10 minutes prior to surgery start (Syringe A). 45 minutes before expected extubation patients will receive morphine 0.15-0.2 mg/kg ideal bodyweight (syringe B).
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Methadone — The dosage administered differ in regards to age and tolerance to opioids:
  0.2 mg/kg: all patients <65 years of age and all patients tolerant to opioids (defined as treatment with opioids (at least the last 7days) exceeding 60 oral morphine milligram equivalents daily.
  0.15 mg/kg: Opioid naive patients > 65 years of age.
  Arms: Methadone, end of surgery; Methadone, induction
Drug: Morphine — The dosage administered differ in regards to age and tolerance to opioids:
  0.2 mg/kg: all patients <65 years of age and all patients tolerant to opioids (defined as treatment with opioids (at least the last 7days) exceeding 60 oral morphine milligram equivalents daily.
  0.15 mg/kg: Opioid naive patients > 65 years of age.
  Arms: Morphine

SUMMARY:
A prospective double-blind, randomized controlled trial investigating the effect of a single-dose of intraoperative methadone in patients undergoing spinal fusion.

DETAILED DESCRIPTION:
During early recovery after surgery, intravenous opioids are typically administered to control the pain, either as intermittent bolus administration by nursing staff or by a patient-controlled analgesia device. Unfortunately, repeated doses or boluses of shorter-acting opioids, such as morphine, oxycodone and fentanyl, result in fluctuating blood concentrations, with the inherent risk of only relatively brief periods of adequate pain relief. Moreover, the use of shorter-acting opioids increases the risk of opioid-associated side effects, such as sedation, nausea and vomiting. An alternative approach to the postoperative use of shorter-acting opioids is therefore called for.

In this respect, methadone is an opioid with unique pharmacological properties that may be advantageous when applied intraoperatively. A single-dose of this long acting opioid could provide a stable analgesia and potentially reduce the need for shorter-acting opioids

Method:

150 patients will be included in an investigator-initiated, prospective, randomised, double-blind, controlled trial with three arms: intervention arm 1 (methadone administered at induction 0.15-0.2 mg/kg ideal body weight), Intervention arm 2 (methadone administered in the end of surgery 0.15-0.2 mg/kg ideal body weight), Control arm (morphine administered in the end of surgery 0.15-0.2 mg/kg ideal body weight).

The study will be GCP-monitored, and is approved by the Danish Health and Medicines Authority (2020103115) and the Central Denmark Region Committees on Health Research Ethics (1-10-72-278-20).

Objective The aim of this study is to investigate the effect of a single dose of intravenous intraoperative methadone on postoperative opioid consumption, pain and side effects in patients scheduled for spinal fusion surgery. A single dose of intravenous intraoperative morphine will be used as an active comparator.

Hypothesis

* Intravenous perioperative methadone reduces opioid consumption (oral cumulative equivalent dose) by 50% during the first 24 postoperative hours compared to intravenous morphine(primary outcome).
* Methadone reduces opioid consumption the first 6 postoperative hours compared to intravenous morphine
* Methadone reduces pain in the affected areas at rest and during coughing(1-72 hours after extubation) compared to intravenous morphine
* Methadone increases patient satisfaction with pain management during the first 24 postoperative hours compared to intravenous morphine on a Numerical Rating Scale (NRS) from 0 to 10, where 0 is unsatisfied and 10 is satisfied
* The effects of methadone is attenuated when administered prior to surgical incision compared to administration in the end of surgery
* The frequency of opioid-related side effects is similar in the groups compared.

ELIGIBILITY:
Inclusion Criteria:

- All patients (≥18 years ≤85) scheduled for elective spinal fusion surgery are screened for inclusion.

Exclusion Criteria:

* Allergy to study drugs
* American Society of Anaesthesiologists (ASA) physical status IV or V
* Prolonged QTc-interval assessed by electrocardiogram(> 440 milliseconds)
* Inability to provide informed consent
* Severe respiratory insufficiency(Oxygen treatment at home)
* Known or clinical signs of heart failure (Ejection Fraction <30%)
* Acute alcohol intoxication/delirium tremens
* Known or clinical signs of increased intracranial pressure
* Acute liver disease
* Acute abdominal pain
* Known or clinical signs of severe liver dysfunction (cirrhosis, inflammation/hepatitis or liver malignancies)
* Known or clinical signs of severe kidney insufficiency(eGFR<30)
* Pregnancy: women of childbearing potential will be tested with serum-HCG prior to surgery, unless the woman is using a birth control method that may be considered as highly effective (based on CTFG 'recommendations related to contraception and pregnancy testing in clinical trials'). Women of childbearing potential is defined as women between menarche and post-menopausal, unless permanently steril. Post-menopausal is defined as no menses for 12 months without alternative medical cause.
* Breastfeeding mothers
* Existing treatment with a high risk of QTc-interval prolongation
* Existing treatment with opioids (at least the last 7days) exceeding 60 mg morphine equivalents daily
* Planned postoperative treatment with epidural analgesics and/or ketamine infusion
* Treatment with rifampicin
* Spinal fusion surgery over >4vertebral levels
* Spinal fusion surgery due to malignant disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Opioid consumption (mean cumulative MME) | 6 hours
  Opioid consumption within the first 6 hours after extubation
Opioid consumption (mean cumulative MME) | 24 hours
  Opioid consumption within the first 24 hours after extubation

SECONDARY OUTCOMES:
Pain intensity (NRS, 0-10) at rest and coughing | 1-72 hours
  Pain intensity from 0-10 in the affected area at when patient is at rest and coughing at the hours: 1, 3, 6, 24, 48 and 72 after extubation
Patient satisfaction with pain management | 24 hours
  Satisfaction with pain management, measured from 0-10, 24 hours following extubation
Nausea and/or vomiting (PONV) | 6 - 24 hours
  Nausea and/or vomiting (PONV) on a 4 point Likert scale (none/mild/moderate/severe) at 6 and 24 hours.
Readiness to discharge | 2-24 hours
  Time from arrival to readiness for discharge from PACU(hours and minutes),
Level of sedation | 1 hour
  Level of sedation at observation in the PACU (Ramsay Sedation Scale at 1 hour after extubation)
Adverse events | 1-24 hours
  Any adverse events in the PACU
  * Hypoventilation (respiratory rate < 10/minutes)
  * Hypoxemia (peripheral oxygen saturation < 94%)
Given treatment according to patient and investigator | 24 hours
  Patient and investigator are asked to asses which treatment they believe was given
3 months follow-up | 3 months
  Pain (NRS 0-10 in the surgical area and legs (left and right), analgesic consumption (opioids MME and secondary analgesics) and quality ogf life (Eq5D)

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No